CLINICAL TRIAL: NCT01266512
Title: Phase II Study of Concurrent Chemoradiotherapy Using IMRT (With Single Photon Emission Computed Tomography/SPECT-CT to Define Functional Lung Volume and Positron Emission Tomography/PET to Define Gross Tumour Volume/GTV) and Docetaxel-cisplatin (or Carboplatin) Followed by Adjuvant Chemotherapy for Inoperable Stage III Non-small-cell Lung Cancer (NSCLC)
Brief Title: Concurrent Chemoradiotherapy Using Intensity Modulated Radiotherapy (IMRT) & Docetaxel-cisplatin (or Carboplatin) Followed by Adjuvant Chemotherapy for Inoperable Stage III Non-small-cell Lung Cancer
Acronym: C-CRISP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_05158; U1111-1115-3573 (Other: UTN)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Radiotherapy, Intensity-Modulated; Cisplatin

ARMS (1):
- IMRT & docetaxel-cisplatin (Experimental): Concurrent chemo-RT:
  Radiotherapy: IMRT - Docetaxel 20mg/m2 + cisplatin 20mg/m2 weekly for 6 weeks -
  Resting period: 2 weeks -
  Adjuvant chemotherapy: Q3W for 2 cycles Docetaxel 35 mg/m² IV infusion for 1 hour on D1&8 - Cisplatin 35 mg/m² on D1&8 -
  Dexamethasone for a total of 3 doses is to be given at a dose of 4 mg at 12 hours, 1 hour before and 12 hours after docetaxel administration
  Interventions: Drug: DOCETAXEL; Radiation: Intensity Modulated Radiotherapy (IMRT); Drug: CISPLATIN

INTERVENTIONS:
Drug: DOCETAXEL — Pharmaceutical form: docetaxel 20mg or 80 mg concentrate for solution for infusion Route of administration: intravenous
Radiation: Intensity Modulated Radiotherapy (IMRT) — 2 Gy per fraction
Drug: CISPLATIN — Pharmaceutical form: solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

* Response rate (by contrast CT scan)

Secondary Objectives:

* Progression-free survival (PFS)
* Overall survival (OS)

DETAILED DESCRIPTION:
The duration of the study for each patient will include an up to 6-week screening phase, 12 weeks treatment phase (including a resting period of 2 weeks) followed by a long-term follow-up.

ELIGIBILITY:
Inclusion criteria:

* Pathologically proven locally advanced, inoperable, confirmed by PET scan (thorax/ upper abdomen) to be International stage III (2009) NSCLC and without multifocal tumours in the lung
* Disease volume encompassible within a tolerable Planning Target Volume treated to 66 Gy
* FEV1 (Force Expiratory Volume in 1 Second) >1000 ml
* Hemoglobin ≥ 9.0 g/dl
* Absolute neutrophil count (ANC) ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Total bilirubin ≥ 1.5 times the upper limit of normal
* ALT (Alanine Aminotransferase) and AST (Aspartate transaminase) ≤ 2.5 x upper limit of normal (≤ 5 x upper limit of normal for patients with liver derangement)
* ECOG (Eastern Cooperative Oncology Group) PS 0-1

Exclusion criteria:

* Previous treatment with chest radiotherapy, chemotherapy or molecularly targeted agents
* Inadequate lung function (Exercise tolerance less than 1 FOS/Fight of stairs, FEV1 < 1 L/sec, or raised pCO2)
* History of hypersensitivity or contraindication to the study drugs or pre-medications or products formulated in polysorbate 80
* Pregnant or breast-feeding women, or women with child-bearing potential who are not following an effective method of contraception and/or who are unwilling or unable to be tested for pregnancy (either by serum or urine pregnancy test before study entry
* Participation in a clinical trial with any investigational drug used and within 30 days prior to study entry

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response rate (by contrast CT scan) | 12 weeks after completion of adjuvant chemotherapy or within 4 weeks after premature study discontinuation

SECONDARY OUTCOMES:
Progression Free survival (PFS) | Day 1 of treatment to the date of objective disease progression
Overall survival (OS) | Day 1 of treatment to the date of death due to any cause
Adverse events (including oesophageal and pulmonary toxicities) | Informed consent signature up to 12 weeks after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong